CLINICAL TRIAL: NCT04236557
Title: Individualized Music Playlist Based on ISO-Principle for De-escalating Agitation of People Living With Dementia: A Randomized Controlled Feasibility Study
Brief Title: Individualized Music Playlist Based on ISO-Principle for De-escalating Agitation of People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Daphne Cheung, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20190731001
Record Dates: First submitted 2019-12-06; First posted 2020-01-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dementia
Keywords: Music; Agitation; Dementia; De-escalation
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Music listening
- Wait-list Control (Placebo Comparator)
  Interventions: Behavioral: Audio Book Listening

INTERVENTIONS:
Behavioral: Music listening — Other than usual care, subjects will listen to a 30-min individualized playlists with preferred music genres sequenced by a registered music therapist according to the ISO-Principle when agitated.
  Arms: Intervention
Behavioral: Audio Book Listening — Other than usual care, subjects will listen to to a 30-min audio-script of book reading in Cantonese (a common dialect in Hong Kong being spoken by most people) when agitated.
  Arms: Wait-list Control

SUMMARY:
Abstract:

Agitation is exhibited by almost every dementia patient during the course of illness, and that leads to detrimental consequences on both patients and caregivers. Listening to preferred music is found useful in reducing the agitation frequency of people with dementia. However, the music intervention is usually provided regularly and the music psychotherapy ISO-Principle is ignored in published studies. The ISO-Principle that commonly adopted in music therapy using live-music, suggests that characteristics of music being played (e.g. tempo, melody and lyrics) should match with the current state (e.g. manic/depressive) of the client, and gradually modify these characteristics to the desired state. This randomized feasibility trial aims to evaluate the feasibility of using individualized music playlist with the music genres sequenced according to the ISO-Principle, for de-escalating agitation of people with dementia, and provide preliminary evidence on efficacy.

Eighty-four nursing home residents with agitation will be randomly allocated into music listening or control groups. Acceptability, implementation and practicality, as well as efficacy (in terms of agitation intensity, stress and mood states before and after the de-escalating music intervention or control condition; and occurrence of agitation and other behavioural and psychological symptoms of dementia before and after the 6-week observation period).

Feasibility indicators will be reported descriptively. The efficacy of (1) music listening in de-escalating symptoms and (2) reducing occurrence frequency of symptoms after 6 weeks, will be analysed with Generalized Estimating Equation. If the findings are positive, the intervention have a great potential to be adopted as the gold standard of care in the nursing homes to solve a common yet detrimental clinical problem.

DETAILED DESCRIPTION:
1. Aims and objectives:

   This study is to evaluate the feasibility of the individualized music playlist based on ISO-Principle for de-escalating agitation of nursing home residents living with dementia.

   Objectives are as below:
   1. To evaluate the feasibility of the intervention in terms of recruitment, retention, and acceptability.
   2. To examine the preliminary effects of the intervention on participants' agitation, stress and emotion as compared to control group.
   3. To evaluate suitability of outcome assessment instruments.
2. Methods:

   1. Design:

      * A two arms randomized controlled feasibility trial.
   2. Participants and setting:

      * The study participants will be recruited from participating residential care homes for the elderly in Hong Kong.
   3. Intervention group

      * Will receive usual care and a 30-minute personalized playlist with the preferred music sequenced according to ISO-Principle will be provided when the participant become agitated during the 6-week project period.
   4. Control group

      * Will receive usual care and a 30-minute audio recording of book reading wen the participant become agitated during the 6-week project period. They will receive a personalized playlist with the preferred music sequenced according to ISO-Principle when all the data collection is done.
   5. Outcomes:

      * recruitment rate, attrition rate, acceptability (field observation, comments from staffs), practicality (adherence to the intervention protocol), and any adverse reactions.
      * agitation severity (Behavioural Activity Rating Scale, Positive and Negative Syndrome Scale Excited Component), heart rate, emotional states (Mood scales derived from DSM-V), before and after listening to the playlist
      * agitation frequency (Cohen-Mansfield Agitation Inventory) and behavioral and psychological symptoms of dementia frequency (Neuropsychiatric Inventory- Questionnaire), at baseline and after 6 weeks
   6. Sample size:

      * 84 participants
   7. Randomization:

      * Participants will be randomly assigned to either intervention or control group at 1:1 ratio.
   8. Data analysis strategies:

      * Descriptive statistics will be used to report the feasibility indicators.
      * The treatment effect on agitation intensity, stress and mood as compared to control group before and after listening to music or control condition for 30 minutes during agitated state, will be analysed using Generalized Estimating Equation (GEE) method.
      * For evaluating the efficacy of music listening in reducing the occurrence frequency of agitation and other behavioural and psychological symptoms of dementia, the scores at baseline and post-intervention (i.e. after 6 weeks) between two groups will be analysed with Mixed ANOVA.
      * Significance level is set at p<.05 with 95% Confidence Interval.
   9. Ethical consideration:

Ethics approval will be obtained from the University before recruiting the participants. Proxies and participants will be informed about the possible risks and benefits of the participation, and it is voluntary and free to withdraw at any time. Procedural consent will be sought too.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents with medical diagnosed of any type of dementia; presented with significant agitation in the past two weeks before recruitment;
* expected to be present in the facility every Monday to Friday during the study period; and
* Aged 60 or above;

Exclusion Criteria:

* Nursing home residents who were admitted to the nursing home for less than 3 months;
* participating in other studies or experimental therapies, or blinded treatments;
* those with comorbid psychiatric illness such as depression, schizophrenia;
* or those with uncorrectable hearing impairment.

Notes:

* Concurrent psychotropic medications over the study period is allowed but any change in the prescriptions will be monitore

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At baseline
  The percentage of eligible participants who finally agreed to join the project
Attrition rate | The 6th week
  The percentage of recruited participant dropped out from the project prematurely
Satisfaction rate | At the end of the 6th week
  Satisfaction of the intervention rated by staff using self-developed rating scale

SECONDARY OUTCOMES:
State of Arousal | During the 6-week study period, before and immediate after listening to the audio when agitated
  To be measured with Behavioural Activity Rating Scale (BARS): a single-item question indicating the condition of the participant in 7-point Likert-scale ranging from 1 - difficult or unable to rouse to 7 - violent, requires restraint. The inter-rater reliability was 0.999 and it is found sensitive in capturing the change of agitation after medication.
Mood States | During the 6-week study period, before and immediate after listening to the audio when agitated
  Mood scales derived from Diagnostic and Statistics Manual - Edition V. It consists of 16 items (8 items for negative mood and positive mood, respectively). with a 0-3 point rating on mood severity.
  the total score of subscale (negative and positive mood) will be calculated. Higher score refers to stronger mood observed.
Agitation frequency | Screening, Baseline, at the end of the project (i.e. the 6th week)
  Cohen-Mansfield Agitation Inventory (CMAI) will be used.
  The CMAI is a caregivers' rating questionnaire consisting of 29 agitated behaviors, each rated on a 7-point scale of frequency. Ratings pertain to the two weeks preceding the administration of the CMAI.
  total score of sub-scale of three factors (Aggressive behaviour, physical non-agggressive behviour, and verbal agitted behaviours) will be calculated. A higher score means more frequent agitation.
Behavioural and psychological symptoms of dementia frequency | Screening, Baseline, at the end of the project (i.e. the 6th week)
  The behavioural and psychological symptoms of dementia frequency will be assessed with Neuropsychiatric Inventory Questionnaire (NPI-Q).
  It consists of 12 items covering the following domains: Hallucinations, Delusions, Agitation/aggression, Dysphoria/depression, Anxiety, Irritability, Disinhibition, Euphoria, Apathy, Aberrant motor behavior, Sleep and night-time behavior change, and Appetite and eating change. Each NPI-Q item is rated by the caregiver as 0-3 points according to levels of increasing severity and the score maximums are determined by multiplying the number of items by 3.
Heart rate | Continuously during the 6-week study period
  Will be measured with wearable sensor
Agitation Intensity | During the 6-week study period, before and immediate after listening to the audio when agitated
  To be measured with Positive and Negative Syndrome Scale Excited Component (PANSS-EC). The PANSS-EC consists of 5 items: excitement, tension, hostility, uncooperativeness, and poor impulse control. The 5 items from the PANSS-EC are rated from 1 (not present) to 7 (extremely severe); scores range from 5 to 35; mean scores ≥ 20 clinically correspond to severe agitation. This set of items detects differences between drug and placebo when evaluating acute agitation and aggression in psychiatric patients [5,7-10] with different psychiatric pathologies.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Sze Ki Cheung, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Cummings J, Mintzer J, Brodaty H, Sano M, Banerjee S, Devanand DP, Gauthier S, Howard R, Lanctot K, Lyketsos CG, Peskind E, Porsteinsson AP, Reich E, Sampaio C, Steffens D, Wortmann M, Zhong K; International Psychogeriatric Association. Agitation in cognitive disorders: International Psychogeriatric Association provisional consensus clinical and research definition. Int Psychogeriatr. 2015 Jan;27(1):7-17. doi: 10.1017/S1041610214001963. Epub 2014 Oct 14. PMID 25311499
- [Background] Palm R, Sorg CGG, Strobel A, Gerritsen DL, Holle B. Severe Agitation in Dementia: An Explorative Secondary Data Analysis on the Prevalence and Associated Factors in Nursing Home Residents. J Alzheimers Dis. 2018;66(4):1463-1470. doi: 10.3233/JAD-180647. PMID 30412491
- [Background] Brimelow RE, Wollin JA, Byrne GJ, Dissanayaka NN. Prescribing of psychotropic drugs and indicators for use in residential aged care and residents with dementia. Int Psychogeriatr. 2019 Jun;31(6):837-847. doi: 10.1017/S1041610218001229. Epub 2018 Nov 20. PMID 30457077
- [Background] Hofmann H, Hahn S. Characteristics of nursing home residents and physical restraint: a systematic literature review. J Clin Nurs. 2014 Nov;23(21-22):3012-24. doi: 10.1111/jocn.12384. Epub 2013 Oct 11. PMID 24125061
- [Background] Cheng ST. Dementia Caregiver Burden: a Research Update and Critical Analysis. Curr Psychiatry Rep. 2017 Aug 10;19(9):64. doi: 10.1007/s11920-017-0818-2. PMID 28795386
- [Background] Zwijsen SA, Kabboord A, Eefsting JA, Hertogh CM, Pot AM, Gerritsen DL, Smalbrugge M. Nurses in distress? An explorative study into the relation between distress and individual neuropsychiatric symptoms of people with dementia in nursing homes. Int J Geriatr Psychiatry. 2014 Apr;29(4):384-91. doi: 10.1002/gps.4014. Epub 2013 Aug 20. PMID 23963653
- [Background] Morris S, Patel N, Baio G, Kelly L, Lewis-Holmes E, Omar RZ, Katona C, Cooper C, Livingston G. Monetary costs of agitation in older adults with Alzheimer's disease in the UK: prospective cohort study. BMJ Open. 2015 Mar 13;5(3):e007382. doi: 10.1136/bmjopen-2014-007382. PMID 25770235
- [Background] Dementia: Assessment, management and support for people living with dementia and their carers. London: National Institute for Health and Care Excellence (NICE); 2018 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK513207/ PMID 30011160
- [Background] Azermai M, Petrovic M, Elseviers MM, Bourgeois J, Van Bortel LM, Vander Stichele RH. Systematic appraisal of dementia guidelines for the management of behavioural and psychological symptoms. Ageing Res Rev. 2012 Jan;11(1):78-86. doi: 10.1016/j.arr.2011.07.002. Epub 2011 Aug 10. PMID 21856452
- [Background] Livingston G, Kelly L, Lewis-Holmes E, Baio G, Morris S, Patel N, Omar RZ, Katona C, Cooper C. Non-pharmacological interventions for agitation in dementia: systematic review of randomised controlled trials. Br J Psychiatry. 2014 Dec;205(6):436-42. doi: 10.1192/bjp.bp.113.141119. PMID 25452601
- [Background] van der Steen JT, Smaling HJ, van der Wouden JC, Bruinsma MS, Scholten RJ, Vink AC. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2018 Jul 23;7(7):CD003477. doi: 10.1002/14651858.CD003477.pub4. PMID 30033623
- [Background] Pedersen SKA, Andersen PN, Lugo RG, Andreassen M, Sutterlin S. Effects of Music on Agitation in Dementia: A Meta-Analysis. Front Psychol. 2017 May 16;8:742. doi: 10.3389/fpsyg.2017.00742. eCollection 2017. PMID 28559865
- [Background] Jacobsen JH, Stelzer J, Fritz TH, Chetelat G, La Joie R, Turner R. Why musical memory can be preserved in advanced Alzheimer's disease. Brain. 2015 Aug;138(Pt 8):2438-50. doi: 10.1093/brain/awv135. Epub 2015 Jun 3. PMID 26041611
- [Background] Tsoi KKF, Chan JYC, Ng YM, Lee MMY, Kwok TCY, Wong SYS. Receptive Music Therapy Is More Effective than Interactive Music Therapy to Relieve Behavioral and Psychological Symptoms of Dementia: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2018 Jul;19(7):568-576.e3. doi: 10.1016/j.jamda.2017.12.009. Epub 2018 Feb 1. PMID 29396186
- [Background] Vasionyte I, Madison G. Musical intervention for patients with dementia: a meta-analysis. J Clin Nurs. 2013 May;22(9-10):1203-16. doi: 10.1111/jocn.12166. PMID 23574287
- [Background] Cheung DSK, Lai CKY, Wong FKY, Leung MCP. Is music-with-movement intervention better than music listening and social activities in alleviating agitation of people with moderate dementia? A randomized controlled trial. Dementia (London). 2020 Jul;19(5):1413-1425. doi: 10.1177/1471301218800195. Epub 2018 Sep 20. PMID 30235949
- [Background] Gaviola MA, Inder KJ, Dilworth S, Holliday EG, Higgins I. Impact of individualised music listening intervention on persons with dementia: A systematic review of randomised controlled trials. Australas J Ageing. 2020 Mar;39(1):10-20. doi: 10.1111/ajag.12642. Epub 2019 Mar 26. PMID 30912616
- [Background] Music & Memory. Impact report. New York.: Music & Memory;2017.
- [Background] Garrido S, Dunne L, Chang E, Perz J, Stevens CJ, Haertsch M. The Use of Music Playlists for People with Dementia: A Critical Synthesis. J Alzheimers Dis. 2017;60(3):1129-1142. doi: 10.3233/JAD-170612. PMID 28984606
- [Background] Gerdner LA. Individualized music for dementia: Evolution and application of evidence-based protocol. World J Psychiatry. 2012 Apr 22;2(2):26-32. doi: 10.5498/wjp.v2.i2.26. PMID 24175165
- [Background] McDermott O, Crellin N, Ridder HM, Orrell M. Music therapy in dementia: a narrative synthesis systematic review. Int J Geriatr Psychiatry. 2013 Aug;28(8):781-94. doi: 10.1002/gps.3895. Epub 2012 Oct 18. PMID 23080214
- [Background] Thoma MV, Zemp M, Kreienbuhl L, Hofer D, Schmidlin PR, Attin T, Ehlert U, Nater UM. Effects of Music Listening on Pre-treatment Anxiety and Stress Levels in a Dental Hygiene Recall Population. Int J Behav Med. 2015 Aug;22(4):498-505. doi: 10.1007/s12529-014-9439-x. PMID 25200448
- [Background] Brown S, Martinez MJ, Parsons LM. Passive music listening spontaneously engages limbic and paralimbic systems. Neuroreport. 2004 Sep 15;15(13):2033-7. doi: 10.1097/00001756-200409150-00008. PMID 15486477
- [Background] Hammar LM, Emami A, Gotell E, Engstrom G. The impact of caregivers' singing on expressions of emotion and resistance during morning care situations in persons with dementia: an intervention in dementia care. J Clin Nurs. 2011 Apr;20(7-8):969-78. doi: 10.1111/j.1365-2702.2010.03386.x. Epub 2011 Feb 10. PMID 21309873
- [Background] Hammar LM, Emami A, Engstrom G, Gotell E. Communicating through caregiver singing during morning care situations in dementia care. Scand J Caring Sci. 2011 Mar;25(1):160-8. doi: 10.1111/j.1471-6712.2010.00806.x. PMID 20573062
- [Background] Ray KD, Fitzsimmons S. Music-assisted bathing: making shower time easier for people with dementia. J Gerontol Nurs. 2014 Feb;40(2):9-13. doi: 10.3928/00989134-20131220-09. Epub 2014 Jan 6. PMID 24550123
- [Background] Wigram T. A comprehensive guide to music therapy : theory, clinical practice, research, and training. London: Jessica Kingsley Publishers; 2002.
- [Background] Altshuler IM. FOUR YEARS'EXPERIENCE WITH MUSIC AS A THERAPEUTIC AGENT AT ELOISE HOSPITAL. American Journal of Psychiatry. 1944;100(7):792-794.
- [Background] Cadwalader A, Orellano S, Tanguay C, Roshan R. The Effects of a Single Session of Music Therapy on the Agitated Behaviors of Patients Receiving Hospice Care. J Palliat Med. 2016 Aug;19(8):870-3. doi: 10.1089/jpm.2015.0503. Epub 2016 Apr 26. PMID 27115462
- [Background] Yuen I, Kwok T. Effectiveness of DementiAbility Methods: The Montessori Way on agitation in long-term care home residents with dementia in Hong Kong. Int J Geriatr Psychiatry. 2019 Sep;34(9):1352-1358. doi: 10.1002/gps.5063. Epub 2019 Mar 1. PMID 30697810
- [Background] Baker RW, Kinon BJ, Maguire GA, Liu H, Hill AL. Effectiveness of rapid initial dose escalation of up to forty milligrams per day of oral olanzapine in acute agitation. J Clin Psychopharmacol. 2003 Aug;23(4):342-8. doi: 10.1097/01.jcp.0000085406.08426.a8. PMID 12920409
- [Background] Kales HC, Gitlin LN, Lyketsos CG. Assessment and management of behavioral and psychological symptoms of dementia. BMJ. 2015 Mar 2;350:h369. doi: 10.1136/bmj.h369. PMID 25731881
- [Background] Swift RH, Harrigan EP, Cappelleri JC, Kramer D, Chandler LP. Validation of the behavioural activity rating scale (BARS): a novel measure of activity in agitated patients. J Psychiatr Res. 2002 Mar-Apr;36(2):87-95. doi: 10.1016/s0022-3956(01)00052-8. PMID 11777497
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Montoya A, Valladares A, Lizan L, San L, Escobar R, Paz S. Validation of the Excited Component of the Positive and Negative Syndrome Scale (PANSS-EC) in a naturalistic sample of 278 patients with acute psychosis and agitation in a psychiatric emergency room. Health Qual Life Outcomes. 2011 Mar 29;9:18. doi: 10.1186/1477-7525-9-18. PMID 21447155
- [Background] Melander C, Martinsson J, Gustafsson S. Measuring Electrodermal Activity to Improve the Identification of Agitation in Individuals with Dementia. Dement Geriatr Cogn Dis Extra. 2017 Dec 6;7(3):430-439. doi: 10.1159/000484890. eCollection 2017 Sep-Dec. PMID 29430245
- [Background] Kikhia B, Stavropoulos TG, Andreadis S, Karvonen N, Kompatsiaris I, Savenstedt S, Pijl M, Melander C. Utilizing a Wristband Sensor to Measure the Stress Level for People with Dementia. Sensors (Basel). 2016 Nov 24;16(12):1989. doi: 10.3390/s16121989. PMID 27886155
- [Background] Schroeder RW, Martin PK, Marsh C, Carr S, Richardson T, Kaur J, Rusk J, Jiwanlal S. An Individualized Music-Based Intervention for Acute Neuropsychiatric Symptoms in Hospitalized Older Adults With Cognitive Impairment: A Prospective, Controlled, Nonrandomized Trial. Gerontol Geriatr Med. 2018 Jun 21;4:2333721418783121. doi: 10.1177/2333721418783121. eCollection 2018 Jan-Dec. PMID 29977982
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Jung SH, Ahn CW. Sample size for a two-group comparison of repeated binary measurements using GEE. Stat Med. 2005 Sep 15;24(17):2583-96. doi: 10.1002/sim.2136. PMID 16118812